CLINICAL TRIAL: NCT05922085
Title: Use of Ultrasound for Early Identification of Patients at Risk of Swallowing Disorders Acquired in the ICU
Acronym: EIDAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PINEDA APPARA 2022
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Patient Under Mechanical Ventilation
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient under mechanical ventilation for at least 48 hours (Experimental)
  Interventions: Other: Ultrasound; Other: nasofibroscopie

INTERVENTIONS:
Other: Ultrasound — performed within 3 hours prior to extubation
Other: nasofibroscopie — performed within 24 to 36 hours after extubation

SUMMARY:
Swallowing disorders (SD) are particularly common after extubation in the ICU and may be associated with an increased risk of lung disease, increased length of hospital stay, and a higher risk of early reintubation. In contrast, early detection of SDs has been shown to be associated with a decrease in these complications. Thus, there is a need for rapid and reliable assessment of SDs in ICU patients before the withdrawal of mechanical ventilation.

Videofluoroscopy (VFS) and nasofibroscopy (NF) are the gold standard examinations for diagnosing SD. However, these two examinations are not feasible in intubated patients.

In this context, ultrasound appears to be a promising alternative to identify patients at risk of SD after extubation. This examination can be performed at the intubated patient's bedside and can be used evaluate the mobility of the structures involved in swallowing. Many studies have already shown the interest of ultrasound in the evaluation of SD but none has focused on intubated patients under respiratory assistance.

The objective of the present study is to evaluate the value of ultrasound in identifying patients at risk of presenting SD after extubation.

This monocentric study will take place in the Intensive Care Unit (ICU) of the Dijon University Hospital. The duration of participation in this research will be equal to the length of stay in the ICU. During their stay, patients will undergo ultrasound and nasofibroscopy. Information on the characteristics of the ICU stay will be collected at discharge.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Major
* On mechanical ventilation for at least 48 hours
* Affiliated to national health insurance

Exclusion Criteria:

Patient:

* Under legal protection (curatorship, guardianship, safeguard of justice)
* Pregnant, parturient or breastfeeding woman
* Refusal to participate by the patient or their proxy (or an immediate family member)
* Cognitive disorders incompatible with the understanding of instructions
* Previously diagnosed swallowing disorders
* With a neurological condition at the origin of the SD (stroke, ALS...)
* Treated for a lesion of the aerodigestive tract (by surgery, radiotherapy or radio-chemotherapy)
* presence of wounds or dressings on the areas to be evaluated that prevent ultrasound measurements
* Patient for whom a decision to limit or stop life support treatments has been taken collegially within the intensive care unit
* With one or more contraindications to performing NF:

  * Anatomical features not compatible with NF: mainly deviation of the nasal septum.
  * Risk of significant otorhinolaryngological bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
rate of swallowing disorders | Within 3 to 24 hours of extubation
  assessed by the Penetration-Aspiration Scale (PAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France